CLINICAL TRIAL: NCT00100750
Title: Gemcitabine and R115777 Combination Therapy for Metastatic Breast Cancer
Brief Title: Tipifarnib and Gemcitabine Hydrochloride in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00114; NCI-2009-00114 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000409695; 2003-0992 (Other: M D Anderson Cancer Center); 7004 (Other: CTEP); P30CA016672 (NIH); N01CM17003 (NIH); N01CM62202 (NIH)
Record Dates: First submitted 2005-01-06; First posted 2005-01-07 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2014-10

CONDITIONS: Recurrent Breast Carcinoma; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; tipifarnib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (gemcitabine hydrochloride, tipifarnib) (Experimental): Patients receive tipifarnib PO BID on days 1-14 and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Gemcitabine Hydrochloride; Drug: Tipifarnib; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdC; dFdCyd
Drug: Tipifarnib — Given PO
  Other Names: R115777; Zarnestra
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I/II trial is studying the side effects and best dose of tipifarnib when given together with gemcitabine hydrochloride and to see how well they work in treating women with breast cancer that has spread to other parts of the body. Tipifarnib is a drug that binds to specific proteins on the tumor cells and then kills these cells. Gemcitabine hydrochloride is a chemotherapy drug that may kill tumor cells by preventing cells from dividing. Giving tipifarnib together with gemcitabine hydrochloride may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the objective response rate of the combination of gemcitabine (gemcitabine hydrochloride) and the farnesyltransferase inhibitor tipifarnib (R115777) in patients with metastatic breast cancer.

II. To evaluate the duration of response, time to disease progression in patients with metastatic breast cancer treated with the combination of gemcitabine and tipifarnib (R115777).

OUTLINE: This is a phase I, dose-escalation study of tipifarnib followed by a phase II study.

Patients receive tipifarnib orally (PO) twice daily (BID) on days 1-14 and gemcitabine hydrochloride intravenously (IV) over 30 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed breast cancer and clinical evidence of metastatic disease
* Patients may have received any number or type of hormonal therapies, either for stage IV disease and/or as adjuvant therapy; patients may have received trastuzumab therapy
* Patients may have received up to 2 prior chemotherapy regimens as therapy for metastatic breast cancer; patients must have recovered from the myelosuppressive effects of prior chemotherapy and all toxicity must have recovered to grade less than or equal to 1
* Concomitant bisphosphonates are allowed for patients with bone metastases
* Localized radiotherapy that does not influence the single evaluable lesion is allowed prior to the initiation of therapy; patients must have recovered from the myelosuppressive effects of previous radiotherapy (at least 4 weeks)
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10 mm with spiral computed tomography (CT) scan
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2 (Karnofsky > 60%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 × institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* There should be a four-week delay between the conclusion of radiation and the start of gemcitabine, provided the acute effects of radiation treatment have resolved

Exclusion Criteria:

* Prior therapy with farnesyltransferase inhibitor or gemcitabine for metastatic breast cancer
* Patients with leptomeningeal disease and/or brain metastasis
* Patients with symptomatic lymphangitic pulmonary metastases
* Patients with peripheral neuropathy greater than or equal to grade 2
* No history of concomitant malignancy except for non-melanoma skin cancer or cervical cancer in situ or other malignancy treated curatively and no evidence of disease for at least five years
* Patients who have had chemotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to tipifarnib (R115777), or imidazole derivatives
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy are excluded from the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-09; Primary Completion 2007-10 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) using the Response Evaluation Criteria in Solid Tumors (RECIST) | Up to 9 years

SECONDARY OUTCOMES:
Time to disease progression using RECIST | Up to 9 years
Incidence of adverse events observed during treatment, graded using the Common Terminology Criteria for Adverse Events version 4.0 | Up to 30 days after completion of study treatment
ORR, by type and extent of prior chemotherapy | Up to 9 years

OTHER OUTCOMES:
Change in serum proteomic analysis | Baseline to up to 9 years

CONTACTS AND LOCATIONS:
Overall Officials: Banu Arun, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States